CLINICAL TRIAL: NCT00753090
Title: Vanguard™ Deep Dish Rotating Platform Knee Clinical Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMETEU.CR.EU13B
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VG DDRP (Experimental): This arm utilizes the Vanguard™ Deep Dish Rotating Platform Knee.
  Interventions: Device: Vanguard™ Deep Dish Rotating Platform Knee
- VG CR (Active Comparator): This arm utilizes the Vanguard™ Cruciate Retaining Knee.
  Interventions: Device: Vanguard™ Cruciate Retaining Knee

INTERVENTIONS:
Device: Vanguard™ Deep Dish Rotating Platform Knee — Total knee replacements with the Vanguard Deep Dish Rotating Platform Knee
  Arms: VG DDRP
Device: Vanguard™ Cruciate Retaining Knee — Total knee replacements with the Vanguard Cruciate Retaining Knee
  Arms: VG CR

SUMMARY:
This study is being conducted on the Vanguard™ Deep Dish Rotating Platform (DD RP) to evaluate the clinical efficacy of the DDRP components.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety and efficacy of Vanguard™ Deep Dish Rotating Platform Knee (mobile bearing knee) as compared to Vanguard Cruciate Retaining Knee (fixed bearing knee). This trial was conducted as the randomised, controlled study.

Implant loosening and polyethylene wear in fixed-bearing knee prostheses were recognized as major causes of late failure. The mobile bearing knee have the theoretical advantages of potentially minimizing the polyethylene wear and reducing implant to bone interface stress in order to reduce the incidence of implant loosening. Therefore, the aims of this study were to prove the Vanguard deep dish rotating platform knee is at least as effective in clinical outcome as the widely used current design of knee replacement and better in long term survivorship.

The efficacy of the device was determined by the relief of pain, restoration of function and range of motion. The durability of device was determined by the absence of revision/removal and radiological integrity. To assess the safety of the device, all post operative complications were recorded either device related or otherwise. Patient satisfaction was determined by answers to patient outcome questionnaires (Oxford Knee Score, WOMAC and Lower Extremity Activity Scale).

Between June 29, 2009 and March 5th 2012, 326 cases were enrolled in the study. In total 117 cases were implanted with the Vanguard fixed bearing cruciate retaining knee; the control arm, and 209 cases were implanted with the Vanguard DDRP. All of these patients fulfilled the inclusion/exclusion criteria. From the 4 participating sites, 2 of them (both located in the Netherlands, Zuyderland Hospital and Bravis Hospital) performed a randomized controlled trial (RCT). In the RCT, 40 cases were assigned to the Trial Arm (Vanguard DDRP), and 51 to the control arm (Vanguard CR). The UK site enrolled cases only in the Vanguard DDRP arm and the French site enrolled in both arms, but non-randomized. Total 326 patients are enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pre-operative Knee Society Score of < 70
* Patients scheduled to undergo primary total knee replacement with any of the following indication: Painful and disabled knee joint resulting from osteoarthritis, Traumatic Arthritis, Rheumatoid Arthritis; One or more compartments are involved
* Need to obtain pain relief and improve function
* Ability and willingness to follow instructions, including control of weight and activity level, and to return for follow-up evaluations
* A good nutritional state of the patient
* Full skeletal maturity of the patient, patients who are at least 18 years of age
* Patients of either sex
* Consent form read, understood, and signed by patient

Exclusion Criteria:

Absolute contraindications include the following diagnoses:

* Patients with a pre-operative Knee Society Score of >= 70
* Infection
* Osteomyelitis
* Previous partial or total prosthetic knee replacement on the operative side
* Patients who are less than 18 years of age
* Sepsis
* Patients who had body mass index >= 40

Relative contraindications include the following factors:

* Uncooperative patient or patient with neurological disorders who are incapable of following directions or who are predictably unwilling to return for follow-up examinations
* Osteoporosis or marked bone loss, which may preclude proper fixation of the prosthesis
* Metabolic disorders, which may impair bone formation
* Osteomalacia
* Distant foci of infections, which may spread to the implant site
* Rapid joint destruction, marked bone loss, or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy, or neuromuscular disease in the affected limb.
* Incomplete or deficient soft tissue surrounding the knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, PhD, Study Director — Zimmer Biomet
Locations (4):
- CHU Lyon Sud, Pierre-Bénite, France
- Netherlands (2):
  - Bravis Ziekenhuis, Roosendaal
  - Zuyderland Medisch Centrum Sittard-Geleen, Sittard
- The Hillingdon Hospital NHS Trust, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who met the criteria were introduced the study by surgeons and got a written information. By the next visit, the surgeons asked if the patients wanted to participate, and if yes, both signed the informed consent. Dutch sites performed randomized controlled trial (RCT). The UK site enrolled the Vanguard DDRP cases only and the French site enrolled both cases without randomization. The UK site was closed after 3 year follow-up, and the French site became unresponsive in 2020.
Groups:
- VG DDRP (Trial Group): This arm utilizes the Vanguard™ Deep Dish Rotating Platform Knee.
- VG CR (Control Group): This arm utilizes the Vanguard™ Cruciate Retaining Knee.
Period: Overall Study
Arm/Group | VG DDRP (Trial Group) | VG CR (Control Group)
Started | 209 | 117
Completed | 41 | 21
Not Completed | 168 | 96
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Death | 17 | 6
Not completed — Study Prosthesis Removed | 12 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Other | 127 | 75

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VG DDRP (Trial Group) | VG CR (Control Group) | Total
Number analyzed (Participants) | 209 | 117 | 326
Age, Continuous [Mean (Full Range); unit: years] | 70.1 [45.0 to 90.0] | 69.0 [18.0 to 87.0] | 69.55 [18.0 to 90.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 67 | 201
  Male | 75 | 50 | 125
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Reason for surgery/indication [Count of Participants; unit: Participants]
  Osteoarthritis | 200 | 115 | 315
  Rheumatoid arthritis | 3 | 2 | 5
  Traumatic arthritis | 1 | 0 | 1
  Other | 5 | 0 | 5
BMI [Mean (Standard Deviation); unit: kg/m²] — Population: Available demographic information is entered.
  kg/m²
    number analyzed (Participants) | 187 | 115 | 302
    (all) | 29.7 (5.5) | 30.0 (4.3) | 29.85 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Knee Society Score
Description: The Knee Society Score (KSS) is a clinician-completed questionnaire and consists of two sub-scores: an Objective score assessing pain, range of motion, anteroposterior and mediolateral stability, along with deductions for higher than normal flexion contracture, extension lag and/or varus/valgus alignment, and a Function score, assessing walking on level ground and walking up and down stairs, along with deductions for support. Each sub-score can range from 0 to 100 points, with higher scores corresponding to better outcomes, classified as Excellent: 80 - 100 points; Good: 70 - 79 points; Fair: 60 - 69 points; Poor: < 60 points.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VG DDRP (Trial Group) | VG CR (Control Group)
Number analyzed (Participants) | 209 | 117
score on a scale
  Objective score | 89.7 (12.0) | 91.8 (9.8)
  Function score | 89.9 (13.9) | 83.2 (21.6)

2. Secondary Outcome: Knee Society Score
Description: as for outcome 1
Time Frame: 6 weeks, 6 months, annually until all available study patients have completed two-year follow up evaluation and alternating odd years or as needed thereafter up to 10 years
Population: Numbers of participants for both groups are lower than the enrolled number of patients, especially pre-op. This is because leg extension is not being captured for a lot of pre-op cases, and therefore no score could be calculated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VG DDRP (Trial Group) | VG CR (Control Group)
Number analyzed (Participants) | 209 | 117
score on a scale
  Preop (Objective Score): number analyzed (Participants) | 179 | 86
  Preop (Objective Score) | 51.2 (13.7) | 53.2 (15.8)
  6 Week (Objective Score): number analyzed (Participants) | 156 | 80
  6 Week (Objective Score) | 72.4 (19.2) | 77.5 (16.7)
  6 Month (Objective Score): number analyzed (Participants) | 145 | 89
  6 Month (Objective Score) | 81.7 (15.6) | 86.4 (11.1)
  1 Year (Objective Score): number analyzed (Participants) | 124 | 93
  1 Year (Objective Score) | 85.8 (14.8) | 88.9 (10.2)
  2 Year (Objective Score): number analyzed (Participants) | 60 | 74
  2 Year (Objective Score) | 89.7 (12.0) | 91.8 (9.8)
  3 Year (Objective Score): number analyzed (Participants) | 57 | 21
  3 Year (Objective Score) | 85.4 (13.7) | 89.5 (8.5)
  5 Year (Objective Score): number analyzed (Participants) | 108 | 40
  5 Year (Objective Score) | 85.7 (13.8) | 92.6 (6.6)
  7 Year (Objective Score): number analyzed (Participants) | 30 | 19
  7 Year (Objective Score) | 86.8 (12.3) | 90.2 (6.8)
  10 Year (Objective Score): number analyzed (Participants) | 18 | 19
  10 Year (Objective Score) | 87.6 (13.0) | 90.6 (7.6)
  Preop (Function Score): number analyzed (Participants) | 198 | 117
  Preop (Function Score) | 51.9 (17.0) | 55.5 (16.7)
  6 Week (Function Score): number analyzed (Participants) | 165 | 104
  6 Week (Function Score) | 64.1 (19.9) | 62.7 (20.3)
  6 Month (Function Score): number analyzed (Participants) | 167 | 112
  6 Month (Function Score) | 79.8 (18.7) | 78.1 (16.7)
  1 Year (Function Score): number analyzed (Participants) | 131 | 100
  1 Year (Function Score) | 86.6 (17.4) | 84.2 (16.8)
  2 Year (Function Score): number analyzed (Participants) | 60 | 74
  2 Year (Function Score) | 89.9 (13.9) | 83.2 (21.6)
  3 Year (Function Score): number analyzed (Participants) | 62 | 34
  3 Year (Function Score) | 81.3 (22.1) | 86.9 (16.1)
  5 Year (Function Score): number analyzed (Participants) | 114 | 40
  5 Year (Function Score) | 79.8 (25.1) | 90.1 (12.8)
  7 Year (Function Score): number analyzed (Participants) | 38 | 19
  7 Year (Function Score) | 70.5 (24.8) | 67.9 (27.7)
  10 Year (Function Score): number analyzed (Participants) | 21 | 23
  10 Year (Function Score) | 90.0 (23.0) | 88.3 (23.5)

3. Secondary Outcome: Radiographic Evaluation: Total Varus Angle
Description: Assessment of patient x-rays by each site investigator: Total varus angle. This is defined as the sum of the femoral flexion (the angle between the femoral median axis and the tibial median axis) and the tibial angle (the angle between the anatomical axis of the femur and the tibia in the anteroposterior view of the knee joint) minus 180 degrees.
Time Frame: 6 weeks, 6 months, 1, 2, 3, 5, 7, and 10 years postoperative
Population: Note that 7 and 10-years radiographic data is limited, this is because the COVID pandemic was impacting those visits. Therefore, the 7 and 10-years information is limited, and results must be interpreted with care.
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | VG DDRP (Trial Group) | VG CR (Control Group)
Number analyzed (Participants) | 209 | 117
Degree
  6 Weeks Total Valgus Angle: number analyzed (Participants) | 163 | 60
  6 Weeks Total Valgus Angle | 3.1 (3.5) | 3.5 (3.7)
  6 Months Total Valgus Angle: number analyzed (Participants) | 157 | 80
  6 Months Total Valgus Angle | 2.9 (3.7) | 3.9 (3.2)
  1 Year Total Valgus Angle: number analyzed (Participants) | 125 | 72
  1 Year Total Valgus Angle | 3.1 (3.7) | 3.9 (3.3)
  2 Year Total Valgus Angle: number analyzed (Participants) | 52 | 45
  2 Year Total Valgus Angle | 2.9 (3.4) | 3.1 (2.9)
  3 Year Total Valgus Angle: number analyzed (Participants) | 60 | 28
  3 Year Total Valgus Angle | 3.2 (4.1) | 3.4 (3.8)
  5 Year Total Valgus Angle: number analyzed (Participants) | 105 | 40
  5 Year Total Valgus Angle | 2.0 (4.2) | 2.3 (3.2)
  7 Year Total Valgus Angle: number analyzed (Participants) | 29 | 19
  7 Year Total Valgus Angle | -0.7 (4.2) | 3.0 (3.0)
  10 Year Total Valgus Angle: number analyzed (Participants) | 8 | 12
  10 Year Total Valgus Angle | 6.6 (4.1) | 3.4 (3.0)

4. Secondary Outcome: Radiographic Evaluation: Radiolucency
Description: Assessment of patient x-rays by each site investigator: Radiolucency Femoral Radiolucency is defined as the total nr of participants with radiolucency measured on the femur in each of the 7 different zones.
  Tibia AP Radiolucency is defined as total nr of participants with radiolucency in each of the 7 zones measured in the AP view X-ray Tibia lateral Radiolucency defined as total nr of participants with radiolucency in each of the 3 zones in the lateral view X-ray Patella Radiolucency is defined as total nr of participants with radiolucency in each of the 5 zones
Time Frame: 6 weeks, 6 months, 1, 2, 3, 5, 7 and 10 years postoperative
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | VG DDRP (Trial Group) | VG CR (Control Group)
Number analyzed (Participants) | 209 | 117
Participants
  6 Weeks Femoral radiolucency: number analyzed (Participants) | 166 | 60
  6 Weeks Femoral radiolucency | 12 | 0
  6 Weeks Tibial AP radiolucency: number analyzed (Participants) | 166 | 60
  6 Weeks Tibial AP radiolucency | 2 | 2
  6 Weeks Tibial Lateral radiolucency: number analyzed (Participants) | 166 | 60
  6 Weeks Tibial Lateral radiolucency | 3 | 1
  6 Weeks Patella radiolucency: number analyzed (Participants) | 166 | 60
  6 Weeks Patella radiolucency | 0 | 0
  6 Weeks Tibial component migration: number analyzed (Participants) | 164 | 60
  6 Weeks Tibial component migration | 2 | 0
  6 Weeks Femoral component migration: number analyzed (Participants) | 165 | 60
  6 Weeks Femoral component migration | 1 | 0
  6 Months Femoral radiolucency: number analyzed (Participants) | 161 | 80
  6 Months Femoral radiolucency | 16 | 7
  6 Months Tibial AP radiolucency: number analyzed (Participants) | 161 | 80
  6 Months Tibial AP radiolucency | 6 | 8
  6 Months Tibial Lateral radiolucency: number analyzed (Participants) | 161 | 80
  6 Months Tibial Lateral radiolucency | 10 | 8
  6 Months Patella radiolucency: number analyzed (Participants) | 161 | 80
  6 Months Patella radiolucency | 0 | 1
  6 Months Tibial component migration: number analyzed (Participants) | 160 | 78
  6 Months Tibial component migration | 2 | 0
  6 Months Femoral component migration: number analyzed (Participants) | 160 | 78
  6 Months Femoral component migration | 0 | 0
  1 Year Femoral radiolucency: number analyzed (Participants) | 130 | 72
  1 Year Femoral radiolucency | 14 | 6
  1 Year Tibial AP radiolucency: number analyzed (Participants) | 130 | 72
  1 Year Tibial AP radiolucency | 9 | 4
  1 Year Tibial Lateral radiolucency: number analyzed (Participants) | 130 | 72
  1 Year Tibial Lateral radiolucency | 11 | 6
  1 Year Patella radiolucency: number analyzed (Participants) | 130 | 72
  1 Year Patella radiolucency | 3 | 0
  1 Year Tibial component migration: number analyzed (Participants) | 127 | 71
  1 Year Tibial component migration | 1 | 1
  1 Year Femoral component migration: number analyzed (Participants) | 127 | 71
  1 Year Femoral component migration | 0 | 1
  2 Year Femoral radiolucency: number analyzed (Participants) | 53 | 45
  2 Year Femoral radiolucency | 4 | 0
  2 Year Tibial AP radiolucency: number analyzed (Participants) | 53 | 45
  2 Year Tibial AP radiolucency | 4 | 1
  2 Year Tibial Lateral radiolucency: number analyzed (Participants) | 53 | 45
  2 Year Tibial Lateral radiolucency | 2 | 0
  2 Year Patella radiolucency: number analyzed (Participants) | 53 | 45
  2 Year Patella radiolucency | 0 | 0
  2 Year Tibial component migration: number analyzed (Participants) | 52 | 45
  2 Year Tibial component migration | 1 | 1
  2 Year Femoral component migration: number analyzed (Participants) | 52 | 45
  2 Year Femoral component migration | 0 | 0
  3 Year Femoral radiolucency: number analyzed (Participants) | 61 | 28
  3 Year Femoral radiolucency | 11 | 1
  3 Year Tibial AP radiolucency: number analyzed (Participants) | 61 | 28
  3 Year Tibial AP radiolucency | 7 | 0
  3 Year Tibial Lateral radiolucency: number analyzed (Participants) | 61 | 28
  3 Year Tibial Lateral radiolucency | 5 | 0
  3 Year Patella radiolucency: number analyzed (Participants) | 61 | 28
  3 Year Patella radiolucency | 1 | 0
  3 Year Tibial component migration: number analyzed (Participants) | 60 | 28
  3 Year Tibial component migration | 0 | 0
  3 Year Femoral component migration: number analyzed (Participants) | 59 | 28
  3 Year Femoral component migration | 0 | 0
  5 Year Femoral radiolucency: number analyzed (Participants) | 113 | 40
  5 Year Femoral radiolucency | 21 | 0
  5 Year Tibial AP radiolucency: number analyzed (Participants) | 113 | 40
  5 Year Tibial AP radiolucency | 4 | 0
  5 Year Tibial Lateral radiolucency: number analyzed (Participants) | 113 | 40
  5 Year Tibial Lateral radiolucency | 3 | 0
  5 Year Patella radiolucency: number analyzed (Participants) | 113 | 40
  5 Year Patella radiolucency | 2 | 0
  5 Year Tibial component migration: number analyzed (Participants) | 111 | 40
  5 Year Tibial component migration | 3 | 0
  5 Year Femoral component migration: number analyzed (Participants) | 111 | 40
  5 Year Femoral component migration | 3 | 0
  7 Year Femoral radiolucency: number analyzed (Participants) | 31 | 19
  7 Year Femoral radiolucency | 14 | 0
  7 Year Tibial AP radiolucency: number analyzed (Participants) | 31 | 19
  7 Year Tibial AP radiolucency | 7 | 0
  7 Year Tibial Lateral radiolucency: number analyzed (Participants) | 31 | 19
  7 Year Tibial Lateral radiolucency | 5 | 0
  7 Year Patella radiolucency: number analyzed (Participants) | 31 | 19
  7 Year Patella radiolucency | 0 | 0
  7 Year Tibial component migration: number analyzed (Participants) | 31 | 19
  7 Year Tibial component migration | 1 | 0
  7 Year Femoral component migration: number analyzed (Participants) | 31 | 19
  7 Year Femoral component migration | 0 | 0
  10 Year Femoral radiolucency: number analyzed (Participants) | 8 | 12
  10 Year Femoral radiolucency | 0 | 0
  10 Year Tibial AP radiolucency: number analyzed (Participants) | 8 | 12
  10 Year Tibial AP radiolucency | 0 | 0
  10 Year Tibial Lateral radiolucency: number analyzed (Participants) | 8 | 12
  10 Year Tibial Lateral radiolucency | 0 | 0
  10 Year Patella radiolucency: number analyzed (Participants) | 8 | 12
  10 Year Patella radiolucency | 0 | 0
  10 Year Tibial component migration: number analyzed (Participants) | 8 | 12
  10 Year Tibial component migration | 0 | 0
  10 Year Femoral component migration: number analyzed (Participants) | 8 | 12
  10 Year Femoral component migration | 0 | 0

5. Secondary Outcome: Survivorship
Description: implant survival at 10 years post surgery and is presented by the number of cases with the implants unrevised
Time Frame: 10 years
Population: The UK site was closed after 3 year follow-up, and the French site became unresponsive in 2020. This explains the low number of long-term follow-up rate.
Measure: Count of Participants; unit: Participants
Arm/Group | VG DDRP (Trial Group) | VG CR (Control Group)
Number analyzed (Participants) | 209 | 117
Participants | 178 | 114

ADVERSE EVENTS:
Time Frame: All adverse events reported were recorded throughout the participation of the study (Up to 10 years). All adverse events were followed until they have abated, or until a stable situation has been reached.
Description: All adverse events reported spontaneously by the subject or observed by the investigator or his staff were recorded.
  However, the Adverse Event Case Report Form didn't categorize seriousness of the events, therefore, all reported adverse events are presented as SAE's.
Arm/Group | VG DDRP (Trial Group) | VG CR (Control Group)
All-Cause Mortality (participants affected / at risk) | 17/209 | 6/117
Serious Adverse Events (participants affected / at risk) | 111/209 | 14/117
Other Adverse Events (participants affected / at risk) | 0/209 | 0/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VG DDRP (Trial Group) (N=209) | VG CR (Control Group) (N=117)
Calf Edema (Vascular disorders) | 1 (1) | 0 (0)
Cardiovascular (Cardiac disorders) | 3 (3) | 0 (0)
Dermatological (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Dislocation/Subluxation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
DVT (Vascular disorders) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematological (Vascular disorders) | 2 (2) | 0 (0)
Implant Oversized (Surgical and medical procedures) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 5 (5) | 2 (2)
Delayed Wound healing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Loosening (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 14 (16) | 4 (4)
Musculoskeletal (non study joint) (Musculoskeletal and connective tissue disorders) | 32 (40) | 1 (1)
Pain (study Joint) (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Psychological (Psychiatric disorders) | 2 (2) | 0 (0)
Pulmonary Embolism (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Reflex Sympathetic Syndrome (Musculoskeletal and connective tissue disorders) | 12 (12) | 0 (0)
respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
revision of study knee (Musculoskeletal and connective tissue disorders) | 12 (12) | 3 (3)
Traumatic Injury (Musculoskeletal and connective tissue disorders) | 6 (7) | 0 (0)
Traumatic Injury (non study joint) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Neurological (Nervous system disorders) | 0 (0) | 1 (1)
Hematoma (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT00753090/Prot_SAP_000.pdf